CLINICAL TRIAL: NCT06705166
Title: Comparative Analysis of Sarcopenia in Rehabilitation Outcomes Following Femoral Neck Fracture: a Study in Normal Weight and Obese Study Cohort
Status: Not yet recruiting | Type: Observational
Sponsor: Shmuel Harofeh Hospital, Geriatric Medical Center (Other Government)
Responsible Party: Principal Investigator, Nechama Monastyrsky, Hospital deputy director, Shmuel Harofeh Hospital, Geriatric Medical Center
Other Study IDs: SH-122-24
Record Dates: First submitted 2024-11-10; First posted 2024-11-26 (Actual); Last update posted 2024-11-26 (Actual); Status verified 2024-11

CONDITIONS: Sarcopenia in Elderly; Sarcopenic Obesity; Frailty; Femoral Fractures
Keywords: older adults; sarcopenia; obesity; rehabilitation; femoral fractures
MeSH Terms: conditions — Frailty; Femoral Fractures; Sarcopenia; Obesity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Normal weight: Patients 60-85 years old whom Suffered a femoral neck fracture in the last year with normal BMI
- Obese: Patients 60-85 years old whom Suffered a femoral neck fracture in the last year with normal BMI

SUMMARY:
Impact of Obesity on Sarcopenia Prevalence and Severity in Elderly Adults Recovering from Femoral Neck Fractures: A Prospective Study

Introduction Age-related muscle loss, or sarcopenia, which includes reductions in both muscle mass and function, is increasingly recognized as a critical health issue in the elderly. Sarcopenia is associated with frailty, disability, and increased mortality. With its rising prevalence, obesity further complicates aging, leading to a condition termed "sarcopenic obesity" (SO), where sarcopenia coexists with obesity. This combination amplifies risks for physical disability, falls, and fractures in older adults. Although sarcopenia and obesity individually contribute to adverse health outcomes, their combined impact on recovery from hip fractures, particularly femoral neck fractures, is under-researched. Hip fractures severely impact the elderly, with over 40% failing to regain pre-fracture functionality and a mortality rate above 35% within three years post-fracture.

This study aims to assess the impact of obesity on sarcopenia prevalence and severity in older adults recovering from femoral neck fractures, addressing an essential gap in understanding SO's role in post-fracture rehabilitation outcomes.

Objectives

* To evaluate the prevalence and severity of sarcopenia among normal-weight versus obese elderly adults post-femoral neck fracture.
* To investigate the association between sarcopenic obesity and functional recovery.
* To determine whether obesity modifies sarcopenia's impact on rehabilitation outcomes.

Risk-Benefit Statement The study entails minimal risk, as all procedures are non-invasive and consistent with routine rehabilitation practices. The potential benefits include enhanced understanding of sarcopenia's effect on hip fracture recovery, which may inform improved rehabilitation practices. Comprehensive health assessments may also benefit participants' post-fracture care.

Study Design Overview This prospective observational study includes hospitalized elderly patients undergoing rehabilitation post-femoral neck fracture. After obtaining informed consent, participants will complete an initial assessment, including demographic information, medical history, cognitive status, and anthropometric measurements. Blood samples will be collected for biochemical markers.

Stratification and Assessment:

Patients will be categorized into normal-weight and obese groups. Comprehensive assessments, including cognitive function, mobility, frailty, muscle strength, and nutritional status, will establish a baseline for studying sarcopenia and obesity's impact on rehabilitation outcomes.

Population and Criteria:

Sample Size: Up to 300 participants

Inclusion Criteria:

* Age 60-85
* Recent femoral neck fracture (within the past year)
* Ability to provide informed consent

Exclusion Criteria:

* Inability to comply with study requirements
* History of neurodegenerative or psychiatric conditions, recent major surgeries (excluding femoral neck fracture), or conditions affecting muscle metabolism

Procedures:

Baseline Evaluation:

* Cognitive Function: Mini-Mental State Examination (MMSE)
* Anthropometric Measurements: BMI from height and weight
* Functional Independence (FIM): Level of independence in daily activities
* Mobility (Up & Go Test): Indicator of balance and mobility
* Frailty and Muscle Strength: Handgrip strength, SARC-F questionnaire, Muscle Strength and Reflex Assessment (MSRA)
* Nutritional Status: Mini Nutritional Assessment (MNA)
* Laboratory Tests: CRP, calcium, vitamin D, CBC

Post-Rehabilitation Evaluation:

After rehabilitation, participants will repeat baseline assessments to determine changes in sarcopenia severity and functional status.

Unscheduled Visits:

Participants may request evaluations outside the scheduled timeline, documented by the investigator as necessary.

Statistical Analysis

* Descriptive Analysis: Mean and standard deviations for continuous data, frequencies for categorical data.
* Comparative Analysis: Independent t-tests to compare normal-weight and obese groups, dependent t-tests for within-group changes.
* Univariate Analysis: Chi-square or Fisher's exact tests with a significance level of P < 0.05.

Ethics and Confidentiality This study will adhere to the Declaration of Helsinki, ICH-GCP guidelines, and applicable regulations. Informed consent will be obtained from all participants, and confidentiality measures will protect patient privacy, with data limited to authorized personnel and anonymized in reports.

Institutional Review Board (IRB) Approval

IRB approval will be obtained from the Israeli Ministry of Health, following ICH-GCP guidelines. The IRB will oversee the study protocol, consent forms, and all participant materials.

Data Storage and Study Termination

Data will be securely stored, with

DETAILED DESCRIPTION:
INTRODUCTION

The global population of older adults (aged 65 and above) is on the rise. In 2017, this demographic constituted 13% of the world's population, and projections indicate that by 2050, it is expected to reach 2.1 billion people. A significant aspect of human aging involves the gradual reduction of skeletal muscle mass. Numerous prospective studies indicate that muscle mass tends to decrease by around 6% per decade after reaching mid-life. Sarcopenia was considered to be purely loss of muscle (lean) mass of the extremities. In 2010, the European consensus redefined sarcopenia by incorporating the loss of function, specifically in walking speed or grip strength, along with the loss of muscle mass. Since then, several consensus groups have adopted similar definitions, now characterizing sarcopenia as the combination of both functional decline and loss of muscle mass. Sarcopenia is closely associated with frailty, physical disability, hospitalization, osteoporosis, osteoarthritis, and even mortality. Handgrip strength is a frequently employed method for assessing muscle strength, offering a straightforward, reliable, and cost-effective means to identify elderly adults who may be at risk for disability.

Older adults will represent the 20% of the population by 2030 and half of them will suffer from obesity. The prevalence of obesity has reached 30-40% of the population, and there are expectations for its incidence to continue rising in the coming decades. Obesity is linked to over 200 medical complications and poses an elevated risk of morbidity and mortality. It stands as the fifth leading cause of death globally. Obesity is marked by the excessive accumulation of white adipose tissue, not only within typical fat depots but also ectopically, a phenomenon that notably compromises physical function. The human body undergoes substantial changes in composition as age advances. Notably, muscle and bone mass show a progressive decline from the third decade of life, while fat mass tends to increase until around the age of 70. People who suffer from obesity experience weight gain and loss throughout their lives on the background of different diets, it is important to underline that diet-induced weight loss is associated with not only fat, but also muscle and bone losses and may further exacerbate age-related sarcopenia and frailty in older adults. The decline in muscle mass and strength, known as sarcopenia, is very common among older adults with obesity (sarcopenic obesity) and is closely associated with frailty. Sarcopenic obesity emerges as a significant factor contributing to physical disability.

Sarcopenia shares common physio-pathological mechanisms and is frequently linked with a high prevalence of osteoporosis. The introduction of the osteo-sarcopenia concept reflects the intersection of sarcopenia and osteoporosis, contributing to notable functional consequences, including an elevated risk of falls and hip fractures. Hip fractures have a significant impact on the daily lives of individuals aged 65 and above, as more than 40% of those who experience a hip fracture fail to regain the functional status they had before the fracture. Hip fractures are correlated with a substantial prevalence of institutionalization and mortality, with rates exceeding 35% within three years of the incident. Sarcopenia could potentially contribute to the loss of function in individuals who experience hip fractures. The prevalence of sarcopenia in older individuals admitted to acute units with hip fractures ranges from 17% to 37%. Sarcopenia serves as a significant prognostic factor for mortality among older patients admitted to acute units.

One study assessed the effect of sarcopenic obesity on ability to function in women with subacute hip fracture, and found that the presence of obesity did not worsen the negative prognostic role of sarcopenia in the short-term recovery of ability to function after hip fracture in women .Another study reviewed 222 patients who underwent orthopedic surgery and found higher prevalence of sarcopenia and sarcopenic obesity among these patients.

There is relatively limited evidence concerning the impact of sarcopenia on the survival of older individuals with hip fractures admitted to rehabilitation units more over there is no reference to obesity sarcopenia. The exclusion of older individuals from clinical trials often limits the relevance of trial results to clinical practice[35, 36]. Pragmatic studies that enroll real-life older participants become crucial in providing insights applicable to daily clinical practice

Muscle mass The worldwide prevalence of sarcopenia in patients with hip fractures is statistically significant. Despite established therapeutic agents and diagnostic criteria for osteoporosis, there is a lack of clear, practical criteria for diagnosing sarcopenia in the clinical setting. Few studies have reported on the evaluation and treatment of sarcopenia in patients with hip fractures. Additionally, the quality of life for postoperative hip fracture patients could be significantly enhanced through the development of precise assessments for muscle regeneration and rehabilitation.

For patients with hip fractures, diagnosis of sarcopenia is based on diagnostic criteria for acute to chronic health care settings. However, evaluation of physical ability in patients with hip fractures is not possible. Only grip strength can be measured. In addition, while measurement of muscle mass is important for patients with hip fractures, whole-body DEXA imaging before surgery is difficult due to pain and anatomical abnormalities at the fracture site.

This study aims to examine the impact of obesity on sarcopenia prevalence and severity in adults recovering from femoral neck fractures. Addressing a gap in current literature, the research endeavors to provide nuanced insights into the interplay between obesity and sarcopenia, contributing valuable knowledge for optimizing rehabilitation strategies in this patient population.

Risk benefit statement Participation in this study carries minimal risk as all assessments and interventions are non-invasive and routinely conducted in rehabilitation settings. The potential benefits include contributing to advancements in understanding sarcopenia following femoral neck fractures, which may lead to improved rehabilitation strategies. Participants will receive comprehensive health assessments that could enhance their overall post-fracture care. The acquired knowledge may benefit not only the individual but also contribute to the broader field of geriatric orthopedics, potentially influencing future clinical practices and patient outcomes Study Objectives The aim of the current study is to evaluate the differences in sarcopenia outcomes and rehabilitation effectiveness between individuals with normal weight and those classified as obese. This investigation aims to provide crucial insights into the distinct impact of body weight on post-fracture recovery, contributing to a more tailored approach in rehabilitation strategies.

Primary endpoint The primary endpoint of this study is to assess and compare the prevalence and severity of sarcopenia between normal-weight and obese cohorts in adults recovering from femoral neck fractures.

STUDY DESIGN 1.1 Overview of the study design This prospective study focuses on hospitalized rehabilitation patients post-femoral neck fracture. After informed consent, participants undergo a comprehensive initial assessment, including demographic details, medical history, lifestyle habits, fracture information, and cognitive status. Blood samples are collected for various biochemical markers.

Upon initial assessment, patients are stratified into two groups based on body weight: normal weight and obese. Following this stratification, a series of assessments are conducted, encompassing cognitive status (MMSE), anthropometric measurements (BMI), functional independence (FIM), mobility (Up & Go Test), frailty, hand grip strength, sarcopenia likelihood (SARC-F), muscle strength and reflexes (MSRA), and nutritional status (MNA). These assessments aim to provide a thorough evaluation of health and functional status, forming the basis for subsequent analyses on the impact of sarcopenia and obesity on post-fracture recovery.

1.2 Study population 1.2.1 Number of subjects The study population will include up to 300 participants, male and female, aged 60 - 85 years, who have been diagnosed with femoral neck fracture.

1.2.2 Inclusion criteria

* Age between 60-85
* Suffered a femoral neck fracture in the last year.
* Subject willing and able to read, understand and sign an informed consent. 1.2.3 Exclusion criteria
* Inability to comply with the study protocol or understand and sign an informed consent
* Diagnosis of a psychiatric disorder prior to the recent femoral neck.
* Active malignancy
* History of other neurodegenerative diseases including Alzheimer's disease (AD), Parkinson's disease (PD), Lewy Body Dementia (LBD), Frontotemporal dementia (FTD), Multiple sclerosis (MS), Amyotrophic lateral sclerosis (ALS), Creutzfeld Jacob disease (CJD), Multisystem atrophy (MSA), Pseudobulbar palsy (PSP), Corticobasal degeneration (CBD), Wernicke Korsakoff syndrome
* Chronic Inflammatory Disorders:(e.g., rheumatoid arthritis, systemic lupus erythematosus).
* Endocrine Disorders: Individuals with endocrine disorders affecting muscle metabolism (e.g., Cushing's syndrome, hyperthyroidism)
* Recent Major Surgeries: Participants who had undergone major surgeries other than femoral neck fracture within the last six months were excluded
* Severe Cognitive Impairment: e.g., advanced dementia were excluded to ensure reliable participation in assessments and accurate reporting of symptoms related to sarcopenia.

  2 Study procedures. 2.1 Screening and baseline evaluation Upon consent, eligible participants will be invited for baseline evaluation that includes the following procedures. The evaluation will be scheduled for up to 6 weeks following consent.
  1. Demographic, clinical data.
  2. Mini-Mental State Examination (MMSE): Cognitive status will be evaluated using the MMSE, a widely used tool to assess orientation, memory, and other cognitive functions.
  3. Anthropometric Measurements: Weight and height will be recorded to calculate the Body Mass Index (BMI)
  4. Functional Independence Measure (FIM): Assessing basic functions, level of independence in activities of daily living.
  5. Up & Go Mobility Test: This test serves as an indicator of mobility and balance.
  6. Frailty Assessment: Evaluating frailty will involve assessing various physical and functional aspects to gauge the patient's vulnerability and resilience.
  7. Hand Grip Strength: Measuring hand grip strength will provide insights into overall muscle strength and functional capacity.
  8. SARC-F:The SARC-F questionnaire will be administered to assess the likelihood of sarcopenia, focusing on strength, assistance with walking, rising from a chair, climbing stairs, and falls.
  9. MSRA (Muscle Strength and Reflex Assessment): This assessment will involve evaluating muscle strength and reflexes, providing a more detailed understanding of the patient's neuromuscular function.
  10. Mini Nutritional Assessment (MNA):The MNA will be utilized to assess the patient's nutritional status, helping identify individuals at risk of malnutrition.
  11. Lab tests.

      2.2 Post rehabilitation evaluation.

      Upon completion of the rehabilitation period, subjects will undergo a comprehensive assessment to evaluate various health and functional parameters. The following tests will be conducted:
* Blood Tests: chemistry panel, calcium, vitamin D, C-reactive protein (CRP), and CBC
* Functional Independence Measure
* Up & Go Mobility Test
* Calf Circumference
* Mini-Mental State Examination
* Hand Grip Strength
* SARC-F questionnaire
* Muscle Strength and Reflex Assessment
* Mini Nutritional Assessment
* Frailty Assessment
* Anthropometric Measurements

2.3 Unscheduled visits Unscheduled visits may be performed at any time during the study at the subject's request or as deemed necessary by the investigator. The date and reason for the unscheduled visit will be recorded.

2.4 Withdrawal criteria and procedures Subjects will be withdrawn if at any time they decide to withdraw consent or if, in the investigator's opinion, it is in the best interest of the subject to be withdrawn for any reason.

3 Statistical Analysis 3.1 Descriptive Statistics Continuous data will be expressed as means ± standard deviations. The normal distribution for all variables will be tested using the Kolmogorov-Smirnov test. Independent t-tests will be performed to compare variables between the two groups. Dependent t-tests will be performed to compare changes within groups. Categorical data will be expressed in numbers and percentages and be compared by chi-square tests. Univariate analyses will be performed using Chi-Square/Fisher's exact tests (where appropriate) to identify significant variables (P < 0.05)

4 Administration and regulation 4.1 Ethics This study will be conducted in compliance with the Declaration of Helsinki (2008), ICH - GCP guidelines and applicable local regulations.

4.2 Informed Consent The investigator (or designee) will obtain written informed consent from the patient participates in this study after adequate explanation of the aims, methods, objectives, and potential hazards of the study and prior to undertaking any study-related procedures. The investigator must utilize a consent form for documenting written informed consent.

After the subject has had time to read the information and feels that all questions have been satisfactorily answered, they will be asked to sign the informed consent form.

The investigator (or designee) will explain to the subjects that they are completely free to refuse to enter the study or to withdraw from it at any time, without any consequences for their further care and without the need to justify. The investigator will complete the informed consent section of the CRF for each subject.

Each subject will be informed that his/her source medical records may be scrutinized by a QA auditor or an inspector from the regulatory authority, in accordance with applicable regulations, that the investigator will protect any personal information not related to the study, and that these persons are bound by the same confidentiality obligations as the subject's family doctor.

4.3 Confidentiality Patients' anonymity will be strictly maintained and their identities are protected from unauthorized parties. The information is not to be disclosed to any third party (except for medical staff or employees or agents directly involved in the conduct of the study or as required by law).

4.4 Institutional review board (IRB) This protocol and any accompanying material including the informed consent documents to be provided to the subject will be submitted by the investigator to the appropriate IRB according to Israeli Ministry of Health and ICH-GCP requirements. Approval from the IRB must be obtained prior to the study initiation.

4.5 Study termination Investigators reserve the right to terminate the study at any time. In terminating the study, the investigators will ensure that adequate consideration is given to the protection of the subjects' interests.

4.6 Study Files The medical records will be maintained adequately to enable good data storage and later on management. Subject's clinical source documents would include (although not limited to) the following: subject's hospital/clinic/ physician's and nurse's notes, appointment book, original laboratory reports, consultant letters, screening and enrolment log etc.

The investigators must arrange for the retention of the subject identification codes and all study documentation as listed above for 15 years after study termination.

4.7 Adverse Events 4.7.1 Definitions: Adverse event (or adverse experience; AE): Any untoward medical occurrence in a study subject, which does not necessarily have a causal relationship to the study treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom or disease temporally associated with the use of a medical product, whether or not considered related to the medicinal product.

Serious adverse event (SAE): Any untoward medical occurrence that fulfils the above definition of an AE and, in addition, at any dose:

* Results in death
* Is life-threatening
* Results in persistent or significant disability/incapacity
* Requires hospitalization or prolongation of existing hospitalization
* Is a congenital anomaly/birth defect
* Any other important medical event that may not be immediately life threatening or result in death or hospitalization but, according to medical and scientific judgment, may jeopardize the subject or require intervention to prevent one or any other of the outcomes listed above. These events should usually be considered serious.

Note: "life-threatening" refers to any adverse experience in which the subject was at immediate risk of death from the reaction at the time of the AE. It does not refer to a reaction that hypothetically might have caused death if it were more severe.

4.7.2 Assessment of AEs Subjects will be monitored for AEs during the entire study and more particularly, during and after each treatment session by clinical inquiry, clinical observation and (when applicable) by clinical examination. AE information will be documented and all subjects will be questioned about AEs at each visit during the treatment period and at the follow-up visits. AEs will also be recorded whenever spontaneously reported by the subject. Event description, date of onset, intensity, duration, treatment for AE, whether the AE was resolved and probable relationship to the study product will be recorded onto CRFs.

The intensity or severity of the AE will be characterized as:

Mild: AE which is easily tolerated Moderate: AE which is sufficiently discomforting to interfere with daily activity Severe: AE which prevents normal daily activities

An adverse event outcome is classified as follows:

* Recovered: the patient has fully recovered from the adverse event with no residual effects observable
* Recovered with sequelae: the patient has fully recovered from the adverse event with residual effects
* Ongoing: adverse event is still ongoing
* Unknown
* Death Reporting of serious adverse events The investigator must record all serious adverse events regardless of treatment or relationship to investigational product as soon as s/he is informed of the event.

Any SAE which occurs after a patient has entered the study (after signing informed consent), must be reported. The original copy of the serious adverse event form must be kept with the documentation at the site.

Patients who have had an SAE during the treatment period must be followed clinically until all parameters (including laboratory), have either returned to normal, have stabilized or are otherwise explained.

SAEs should be reported by the investigator to competent authorities and ethics committees according to local requirements.

4.8 Financing The study doesn't have funding 4.9 Insurance Coverage by the Shmuel harofeh Medical Center insurance that includes investigator initiated clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Age between 60-85
* Suffered a femoral neck fracture in the last year.
* Subject willing and able to read, understand and sign an informed consent.

Exclusion Criteria:

* Inability to comply with the study protocol or understand and sign an informed consent
* Diagnosis of a psychiatric disorder prior to the recent femoral neck.
* Active malignancy
* History of other neurodegenerative diseases including Alzheimer's disease (AD), Parkinson's disease (PD), Lewy Body Dementia (LBD), Frontotemporal dementia (FTD), Multiple sclerosis (MS), Amyotrophic lateral sclerosis (ALS), Creutzfeld Jacob disease (CJD), Multisystem atrophy (MSA), Pseudobulbar palsy (PSP), Corticobasal degeneration (CBD), Wernicke Korsakoff syndrome
* Chronic Inflammatory Disorders:(e.g., rheumatoid arthritis, systemic lupus erythematosus).
* Endocrine Disorders: Individuals with endocrine disorders affecting muscle metabolism (e.g., Cushing's syndrome, hyperthyroidism)
* Recent Major Surgeries: Participants who had undergone major surgeries other than femoral neck fracture within the last six months

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include up to 300 participants, male and female, aged 60 - 85 years, who have been diagnosed with femoral neck fracture and hospitalized for rehabilitation in Shmuel Harofe geriatric hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2026-01-01 (Estimated)

PRIMARY OUTCOMES:
Sarcopenia screening using the SARC-F questioner | From enrolment to end of the end of rehabilitation, (average 4 weeks)
  Sarcopenia screening using the SARC-F questioner among normal-weight versus obese elderly adults post-femoral neck fracture and comparing it to other tests evaluating patients functional status such as the time up and go, Functional Independence Measure and hand grip and their relation to clinical outcomes such as mortality, length of hospitalization and rehabilitation outcomes. SARC-F is a 5 question sarcopenia screening tool with a score range of 0-10 and sores equal or greater than 4 is predictive of sarcopenia.

IPD SHARING:
Plan to Share IPD: No